CLINICAL TRIAL: NCT04141709
Title: Effektivität Und Toxizität Einer Perkutanen Hochdosierten Strahlentherapie Bei Patienten Mit Oligometastasen Eines Kastrationsresistenten Prostatakarzinoms
Brief Title: Local Ablative Radiotherapy for OLIgoprogressive Castration Resistant Prostate Cancer
Acronym: OLI-CR-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Tobias Hölscher, Principal Investigator, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR - Oli-CR-P - 2018
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Oligometastatic Disease; Prostatic Cancer, Castration-Resistant
Keywords: Oligometastatic Disease; Prostate Cancer; Radiation therapy; Prostatic Cancer, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — Photons

STUDY DESIGN:
Intervention Model Description: 2:1 randomized allocation to intervention (local ablative radiotherapy) or standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local ablative radiotherapy (Experimental): The therapy is performed for all patients in the intervention arm using high-dose radiation therapy, either as conventional fractional irradiation with 2 Gy/fraction up to a total dose of 50 Gy or as hypofractional irradiation with a single dose of 10 Gy up to a total dose of 30 Gy.
  Interventions: Radiation: local ablative radiotherapy
- Observational group (No Intervention): Effectiveness is measured as the rate in patients with PSA progression one year after randomization (defined as PSA nadir after randomization +2 ng/ml).
  There is a 2:1 randomization between intervention and observation group.

INTERVENTIONS:
Radiation: local ablative radiotherapy — Within the scope of the study, irradiation with two irradiation schemes is possible (the scheme applied is recorded in the CRF):
  * Scheme A 3*10 Gy (once a day, 2-3 days a week)
  * Scheme B 25*2 Gy (once a day, 5 days a week) The decision which irradiation scheme (3*10 Gy or 25*2 Gy) to use is made by the treating physician based on the anatomical position, the size of the metastases and the expected normal tissue load. Hypofractionated irradiation in three fractions is only possible if the limit values for the risk organs are adhered to. Radiotherapy should be performed with photons.
  Other Names: Photons
  Arms: local ablative radiotherapy

SUMMARY:
The purpose of this randomized trial is to investigate the efficacy and toxicity of percutaneous high-dose radiotherapy in patients with oligometastases of hormone refractory prostate cancer. The effectiveness will be tested in comparison to an observation group, in which no further therapy is initially given. Treatment can be stereotactically hypofractionated or conventionally fractionated.

DETAILED DESCRIPTION:
This is a monocentric, randomized, prospective Phase II intervention trial. Efficacy is measured as the rate in patients with PSA progression one year after randomization (defined as PSA nadir after randomization +2 ng/ml). There is a 2:1 randomization between intervention and observation group. Patients with PSA progression in the observation group are offered a new diagnosis. This should preferably correspond to the initial diagnosis.

Therapy is performed for all patients in the intervention arm using high dose radiation therapy, either as conventional fractional irradiation with 2 Gy/fraction up to a total dose of 50 Gy or as hypofractional irradiation with a single dose of 10 Gy up to a total dose of 30 Gy.

The decision as to which regimen the patient is to be treated according to is made by the treating physician, taking into account in particular the location of the volume to be irradiated in relation to the organs at risk and any previous irradiation.

ELIGIBILITY:
Indication:

Oligometastases (1-5) in castration-resistant prostate carcinoma

Inclusion Criteria:

* Patient with good general condition (WHO 0-1)
* Histologically confirmed prostate carcinoma
* After definitive local therapy, e.g. radical prostatectomy or definitive radiotherapy (also after neo-adjuvant hormone therapy, after postoperative radiotherapy).
* PSA progression under ongoing androgen deprivation (defined as three consecutive increasing PSA values at intervals of > 4 weeks and testosterone in the castration area <50ng/dl or <1.73nmol/)
* Minimum duration of androgen deprivation 6 months before inclusion in study
* Present complete staging (max. 6 weeks old), preferably by means of PET hybrid imaging with prostate-specific PET tracer
* Imaging detection of individual active or progressive metastases (max. 5, depending on location) that are accessible to local ablative radiotherapy (histological confirmation of the metastases is not required)
* No parallel participation to further clinical therapy trials up to 4 weeks before and after radiation therapy
* Individual case discussion in an interdisciplinary tumor board
* Patient's ability to consent and written consent

Exclusion Criteria:

* Severe concomitant disease that limits further life expectancy to < 5 years according to the physician's assessment.
* PSA > 20ng/ml, testosterone >50 dl or >1,73nmol/l
* visceral metastasis (e.g. lung, liver, brain)
* lack of compliance
* previous taxane-containing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to PSA progression | 12 month after randomization
  Time to PSA progression (defined as PSA nadir after randomization +2ng/ml)

SECONDARY OUTCOMES:
Change of PSA doubling time | 12 month after randomization
  PSA doubling time measured with the last three consecutive PSA values. Change of PSA doubling time compared to value before treatment
Number of patients without detection of new lesions | 12 month after randomization
  Number of patients without detection of new lesions at 12 months
Toxicity (CTCAE 5.0) | 3 and 12 month after therapy
  description of toxicity (CTCAE 5.0) ant 3 and 12 months.
Number of patients who have PSA response | 12 month after randomization
  Number of patients who have a PSA reduction of >50% at 12 months.
Time to tumor-specific systemic therapy after intervention | 12 month after randomization
  Time to tumor-specific systemic therapy after intervention (i.e. chemotherapy)
Number of patients with a limited number of metastases at PSA progression | 12 month after randomization
  Number of patients with a limited number of metastases at PSA progression, compared to patients with multiple metastases. (Arm B only)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hölscher, Dr., Principal Investigator — Radiation Oncology, Technische Universität Dresden
Locations (1):
- Department of Radiotherapy and Radiation Oncology, Faculty of Medicine and University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Saxony, Germany